CLINICAL TRIAL: NCT05629975
Title: Department of Thoracic Surgery, Shanghai Tongji Hospital, School of Medicine, Tongji University, Xincun Rd. 389, Shanghai, 200065, People's Republic of China.
Brief Title: Oral Nutritional Supplements in Treatment of Elderly Mild-to-Moderate COVID-19
Acronym: ONSITEMC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Yongxin Zhou, Doctor, Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SBKT-2022-201
Record Dates: First submitted 2022-11-03; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Nutrition, Healthy
Keywords: Oral nutritional supplements
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to the normal diet in the hospital, patients in the intervention group received a package of nutritional powder in the morning and evening of every day, and each package was diluted with 500 ml of water.
  Each package contained L-arginine (750 mg), methionine (300 mg), glutamine (5 g), plant protein (10 g), vitamin B12 (1 ug), vitamin C (50 mg), vitamin D (2000 IU), vitamin A (300 mg), folic acid (5 mg), omega-3 fatty acid (1 g), zinc (20 mg), magnesium (400 mg), selenium (100 mcg), whole wheat fiber (5 g), carotenoid (3 mg), curcumin supplement (500 mg).
  Probiotics included orally administration of clostridium butyricum& bifidobacterium (500 mg) every day for 7 days.
  Interventions: Dietary Supplement: Oral Nutritional Supplements
- Control group (No Intervention): Patients in the control group received normal diet provided by the hospital.

INTERVENTIONS:
Dietary Supplement: Oral Nutritional Supplements — Each package contained L-arginine (750 mg), methionine (300 mg), glutamine (5 g), plant protein (10 g), vitamin B12 (1 ug), vitamin C (50 mg), vitamin D (2000 IU), vitamin A (300 mg), folic acid (5 mg), omega-3 fatty acid (1 g), zinc (20 mg), magnesium (400 mg), selenium (100 mcg), whole wheat fiber (5 g), carotenoid (3 mg), curcumin supplement (500 mg).
  Probiotics included orally administration of clostridium butyricum& bifidobacterium (500 mg) every day for 7 days.
  Arms: Intervention group

SUMMARY:
The coronavirus disease 2019 (COVID-19) pandemic has seriously threatened public health worldwide. Nutritional supplements may have a positive influence on the recovery of patients with viral infection. This study aimed to assess the influence of oral nutritional supplements (ONSs) on the biochemical parameters of elderly patients with mild-to-moderate COVID-19.

This clinical trial will be conducted on 145 elderly patients with mild-to-moderate COVID-19. Patients in the intervention group (n=74) received nutritional powder (vitamins, minerals, dietary fiber, polyphenols, omega-3, amino acids, and probiotics) for 14 days. Cases in the control group (n=71) took the placebo, except for nutritional powder, and they received the same treatment. Biochemical parameters were measured before and two weeks after intervention.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic has seriously threatened public health worldwide. Nutritional supplements may have a positive influence on the recovery of patients with viral infection. This study aimed to assess the influence of oral nutritional supplements (ONSs) on the biochemical parameters of elderly patients with mild-to-moderate COVID-19.

This clinical trial will be conducted on 145 elderly patients with mild-to-moderate COVID-19. Patients in the intervention group (n=74) received nutritional powder (vitamins, minerals, dietary fiber, polyphenols, omega-3, amino acids, and probiotics) for 14 days. Cases in the control group (n=71) took the placebo, except for nutritional powder, and they received the same treatment. Biochemical parameters were measured before and two weeks after intervention.

After 14 days, patients in the groups will be measured by C-reactive protein (CRP), creatinine (Cr), blood urea nitrogen (BUN), and interleukin-8 (IL-8) ,white blood cell (WBC), red blood cell (RBC), platelet (PLT), neutrophil percentage (NE%), prothrombin time (PT), D-Dimer (DD), blood glucose, sodium (Na+), potassium (K+), aspartate aminotransferase (AST), glutamate pyruvic transaminase (ALT), albumin, calcium (Ca), arterial blood gas (ABG) parameters, and interleukin-10 (IL-10).

ELIGIBILITY:
Inclusion Criteria:

1. COVID-19-positive was confirmed by reverse transcription-polymerase chain reaction (RT-PCR);
2. Mild-to-moderate COVID-19 patients who aged 60-90 years old;
3. Consistency with the indication of enteral nutrition;
4. The time from diagnosis of COVID-19 to hospitalization was less than 24 h.

Exclusion Criteria:

1. Oxygen saturation < 93% or mechanical ventilation was required;
2. Systemic diseases (malignant tumors, autoimmune diseases, liver or kidney diseases);
3. Participation in other clinical trials within 3 months;
4. History of allergy to nutrients in the trial.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
coagulation function and blood cell count (CBC) | 2 weeks
  white blood cell (WBC) count(*109/L)
kidney functions | 2 weeks
  blood urea nitrogen (BUN)(mg/L)
ABG parameters | 2 weeks
  oxygen partial pressure (PO2)(mmHg)
serum electrolytes | 2 weeks
  potassium (K+)(mmol/L)
inflammatory indices | 2 weeks
  interleukin-8 (IL-8)(pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Yongxin Zhou, Dr, Study Chair — Shanghai Tongji Hospital, Tongji University School of Medicine

IPD SHARING:
Plan to Share IPD: No